CLINICAL TRIAL: NCT01378650
Title: A Randomized, Prospective, Placebo-controlled Double-blind, Pilot Study on the Effect of Cilostazol for 4 Weeks in Patients With Chronic Tinnitus
Brief Title: A Study on the Effect of Cilostazol in Patients With Chronic Tinnitus
Acronym: CITI-ESR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jong Woo Chung (Other)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jong Woo Chung, MD, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMC-2010-0800; KCT0000128 (Registry Identifier: Clinical Research Information Service (CRIS))
Record Dates: First submitted 2011-06-21; First posted 2011-06-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Tinnitus
Keywords: Tinnitus; Medication therapy management; Cilostazol; Antiplatelet agents
MeSH Terms: conditions — Tinnitus | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cilostazol group (Experimental): Administration of Cilostazol 100mg twice a day for 4 weeks
  Interventions: Drug: Cilostazol
- Placebo group (Placebo Comparator): placebo drug twice a day for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol — Administration of Cilostazol 100mg twice a day for 4 weeks
  Other Names: Pletaal
  Arms: Cilostazol group
Drug: Placebo — placebo one tablet matching for cilostazol twice a day for 4 weeks.
  Other Names: Placebo matching for cilostazol
  Arms: Placebo group

SUMMARY:
1. Overview of tinnitus Tinnitus is a noisy sound which is perceived without any external sound source. According to the survey of the US, 10-20% of adult have the symptom of tinnitus and 3-5% of tinnitus patients have severe discomfort of daily life. Severe tinnitus can result in psychiatric problems such as depression and anxiety disorders. Enhancement of environmental sound, hearing aids, sound generators, cognitive therapy, transcranial magnetic therapy, and drug therapy have been tried for treatment of tinnitus. Nitric oxide(NO) is a well-known neurotransmitter acting as a vasodilator through regulation of production of cyclic guanosine monophosphate(cGMP) and can be found in various sites of cochlea. It is reported that cGMP enhances activity of protein kinase A (PKA), a mediator of platelet aggregation inhibition and vasodilatation and results in increase of vascular flow.
2. Characteristics of the clinical research drug, cilostazol Cilostazol inhibits phosphodiesterase type 3 (PDE3) selectively and increases amount of cAMP by inhibition of degradation of cyclic adenosine monophosphate(cAMP). cAMP again by increasing the active form of PKA suppress the production of blood clots and increase blood flow by expanding blood vessels. Anti-platelet activity and vasodilatation effect of cilostazol have been used for improvement of diabetic peripheral vascular disorders and suppression of stroke recurrence. Previous studies reported that by increasing the activity of NO and PKA, the blood flow of stria vascularis and cochlear hair cells can be improved. These studies implies that cilostazol, which causes inhibition of PDE3 and increase of PKA, can have a potential effect on improvement of tinnitus by increase of blood flow to peripheral cochlear cells. Thus, we hypothesized that cilostazol, which has been widely used for enhancing peripheral blood flow, can bring improvement of tinnitus by causing better peripheral blood flow of cochlea.
3. The aim of the study We planned this study to validate the assumptions of the background. The aim of our study is whether administration of cilostazol can improve tinnitus in terms of subjective degree of symptoms in chronic tinnitus patients.

DETAILED DESCRIPTION:
1. Clinical research methods

   * Determination of eligibility by history taking, physical examination, pure tone audiometry, speech audiometry, and distortion product otoacoustic emission test.
   * Randomization by random sequence generation
   * Administration : cilostazol 100mg Bid 4 weeks for the study group and placebo tablet Bid 4 weeks for the control group.
   * Evaluation battery: questionnaires (tinnitus handicap inventory, visual analogue scale, Quality of life SF-36)
   * Time of evaluation : pre-administration, 2 weeks after administration, 4 week after administration
   * Monitoring of side effects
2. Evaluation of treatment response - Statistical analysis of scores of questionnaires using SPSS K12.0 (paired t-test for changes of each group and Mann-Whitney U test for comparing the mean scores of two groups)

ELIGIBILITY:
Inclusion Criteria:

* Adults of age over 19
* Unilateral or bilateral tinnitus
* Chronic tinnitus lasting more than 3 months
* Initial visual analogue scale of tinnitus >3

Exclusion Criteria:

* Conductive hearing loss on pure tone audiometry
* Associated other inner ear diseases such as Meniere's disease
* Objective or pulsatile tinnitus
* Contraindication to anti-platelet drug
* Any cardiac disease
* Bleeding tendency and major operation within 3 months
* Breastfeeding
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change of the tinnitus handicap inventory (THI) score | within 2 weeks before administration, 2 weeks after administration, 4 week after administration
  A Questionnaire for assessing subjective discomfort from chronic tinnitus

SECONDARY OUTCOMES:
Changes of Quality of Life (SF-36) score | within 2weeks before administration, 2 weeks after administration, 4 weeks after administration
  A questionnaire for assessing subjective discomfort from chronic tinnitus
Change of the visual analogue scale (VAS) score | within 2 weeks before administration, 2 weeks after administration, 4 week after administration
  A Questionnaire for assessing subjective discomfort from chronic tinnitus

CONTACTS AND LOCATIONS:
Overall Officials: Jong Woo Chung, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Mazurek B, Haupt H, Szczepek AJ, Sandmann J, Gross J, Klapp BF, Kiesewetter H, Kalus U, Stover T, Caffier PP. Evaluation of vardenafil for the treatment of subjective tinnitus: a controlled pilot study. J Negat Results Biomed. 2009 Feb 17;8:3. doi: 10.1186/1477-5751-8-3. PMID 19222841
- [Background] Ye YL, Shi WZ, Zhang WP, Wang ML, Zhou Y, Fang SH, Liu LY, Zhang Q, Yu YP, Wei EQ. Cilostazol, a phosphodiesterase 3 inhibitor, protects mice against acute and late ischemic brain injuries. Eur J Pharmacol. 2007 Feb 14;557(1):23-31. doi: 10.1016/j.ejphar.2006.11.003. Epub 2006 Nov 10. PMID 17161838
- See also: Clinical Research Information Service (CRIS) — https://cris.nih.go.kr/cris/index.jsp
- See also: Institutional Review Board of Asan Medical Center — http://crc.amc.seoul.kr